CLINICAL TRIAL: NCT00006191
Title: Effects of Levetiracetam on Cortical Excitability in Humans
Brief Title: Effect of Levetiracetam on Brain Excitability
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000207; 00-N-0207
Record Dates: First submitted 2000-08-29; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-08

CONDITIONS: Healthy; Myoclonic Epilepsy
Keywords: Antiepileptic Drugs; Motor Cortex; Myoclonus; Healthy Volunteer
MeSH Terms: conditions — Epilepsies, Myoclonic; Myoclonus

SUMMARY:
This study will examine the effect of the newly developed anti-epileptic drug, levetiracetam, on excitability of the cortex (surface layer) of the brain. Levetiracetam works differently from other anti-seizure drugs, but its mechanism is not well understood. This study may provide insight into a new protection mechanism against seizures as well as the effect of the drug on cortical excitability.

Healthy normal volunteers 18 years of age and older may be eligible for this study. Candidates will have a medical history taken and undergo physical and neurological examinations.

Participants will undergo two different procedures in four separate sessions. One procedure (cortical excitability) involves taking either levetiracetam or placebo (a look-alike inactive substance) and having transcranial magnetic stimulation (TMS). The other procedure (pinch-training related changes) involves taking levetiracetam or placebo, doing a motor exercise called pinch training, and having transcranial magnetic stimulation. For TMS, a very brief electrical current is passed through an insulated coil wire placed on the scalp. The magnetic pulse travels through the scalp and skull, causing small electrical currents in the cortex that may cause muscle, hand, or arm twitching or it may affect movements or reflexes. During the study, subjects may be asked to make movements, do simple tasks or tense muscles. Electrical activity of the muscles will be recorded using electrodes taped to the skin over the muscle. For the pinch training, the subject makes a brief, brisk pinch after each beat of a metronome every two seconds and then completely relaxes the hand until the next beat.

Subjects will be tested on four different days at least 72 hours apart. Each session will last about 3 to 4 hours.

Approximate schedule for cortical excitability testing:

TMS (study 1)

Take levetiracetam or placebo

TMS (study 2) < 60 minutes after drug or placebo

TMS (study 3) < 120 minutes after drug or placebo

Approximate schedule for pinch-training related changes:

Take levetiracetam or placebo

TMS and pinch power measurement < 60 minutes after drug or placebo

Pinch training for 30 minutes

TMS and pinch power measurement

Sample schedule:

Session 1 < LTC and cortical excitability testing

Session 2 < Placebo and cortical excitability testing

Session 3 < LTC and pinch-training related changes

Session 4 < Placebo and pinch-training related changes

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of newly developed antiepileptic drug, levetiracetam, on cortical excitability in humans. This drug may be useful in patients with myoclonus, and its mode of action is not well understood. We plan to determine if oral administration of levetiracetam in therapeutic dosage alters cortical excitability measured by transcranial magnetic stimulation as well as long-term potentiation measured by pinching practice in humans.

ELIGIBILITY:
This study will be done on normal volunteers.

Subjects will be adults older than age 18.

No development of a serious medical condition.

Compliance with protocol evaluations or examinations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14
Dates: Start 2000-08; Study Completion 2001-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bialer M, Johannessen SI, Kupferberg HJ, Levy RH, Loiseau P, Perucca E. Progress report on new antiepileptic drugs: a summary of the fourth Eilat conference (EILAT IV). Epilepsy Res. 1999 Mar;34(1):1-41. doi: 10.1016/s0920-1211(98)00108-9. PMID 10194110
- [Background] Wulfert E, Hanin I, Verloes R. Facilitation of calcium-dependent cholinergic function by ucb L059, a new "second generation" nootropic agent. Psychopharmacol Bull. 1989;25(3):498-502. PMID 2626523
- [Background] Loscher W, Honack D. Profile of ucb L059, a novel anticonvulsant drug, in models of partial and generalized epilepsy in mice and rats. Eur J Pharmacol. 1993 Mar 2;232(2-3):147-58. doi: 10.1016/0014-2999(93)90768-d. PMID 8467854